CLINICAL TRIAL: NCT00784329
Title: Pilot Study To Evaluate Optical Frequency Domain Imaging For Diagnosis Of Central Airway Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Lahey Clinic (Other)
Collaborators: Massachusetts General Hospital (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2008-031
Record Dates: First submitted 2008-10-31; First posted 2008-11-03 (Estimated); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Squamous Cell Lung Cancer; Lung Cancer; Pulmonary Disease
Keywords: Lung Cancer; Squamous Cell Lung Cancer; Bronchial carcinoma in situ; Central Airway Diseases
MeSH Terms: conditions — Lung Neoplasms; Lung Diseases | interventions — Drug Delivery Systems; Bronchoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Optical Frequency Domain Imaging (Experimental): Optical Frequency Domain Imaging System used during Lung and Bronchial biopsies to detect cancerous tissue. Tissue imaging results will be compared to tissue biopsy results.
  Interventions: Device: Optical Frequency Domain Imaging (OFDI) System

INTERVENTIONS:
Device: Optical Frequency Domain Imaging (OFDI) System — Optical Frequency Domain Imaging(OFDI)System. Additional biopsy obtained from regions of normal appearing tissue. Up to an additional 20 minutes to standard Bronchoscopy
  Other Names: Lung tissue biopsy; Tissue imaging by Optical Frequency; Bronchoscopy

SUMMARY:
To evaluate the potential of a new imaging device, termed Optical Frequency Domain Imaging (OFDI), in the early diagnosing of pulmonary malignancies in the central airways.

DETAILED DESCRIPTION:
This study will evaluate the potential of a new imaging device, the Optical Frequency Domain Imaging (OFDI) for imaging pulmonary malignancy in the central airways.

The prevalence and high mortality rate associated with Lung Squamous Cell Carcinoma and the lack of any widely accepted screening and surveillance tools, highlights the need for new imaging paradigms that will ultimately lead to a reduction in patient mortality.

Bronchial carcinoma in-situ will progress to invasive cancer in over 40% of individuals, and although the progression occurs over a long period of time, the majority of carcinomas are detected in the later stages of disease development, offering patients only a very slim chance of cure. Although, significant effort in the development of screening paradigms for the detection of lung cancer in the central airway has been made, to date there is still no widely accepted and validated approach. Optical Frequency Domain Imaging (OFDI) is a recent derivative of optical coherence tomography (OCT). As in OCT, OFDI is an interferometric ranging technique that can roughly be considered to be an optical analogue of ultrasound imaging and can provide tomographic images of tissue at resolutions comparable with architectural histology. The long term goal of this study is to use OFDI to screen the airways with the hope of detecting Squamous Cell Carcinoma at an earlier more curable stage.

Standard of care bronchoscopy preparation and procedures to be followed, with moderate sedation, pulse oximetry and blood pressure monitoring as per department protocol. A combination of currently approved bronchoscopy techniques including stand white light bronchoscopy, autofluorescence bronchoscopy, and narrow band imaging will be used to assess the airways.

Bronchial regions of interest (ROI's)suspected to be premalignant or malignant, identified during the bronchoscopy procedure, will be imaged using the OFDI system and catheter before biopsy is done. It is anticipated to obtain a minimum of 3 OFDI-biopsy correlated pairs from each study participant. An additional OFDI image and biopsy will be obtained from region's of normal interest (ROI's). It is expected that the experimental procedure will add less than 10 minutes to the total length of the bronchoscopy procedure, but a stopping rule will be instituted to ensure that the experimental procedure does not exceed 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing bronchoscopy for known or suspected pulmonary malignancy in the central airways
* Patients must be over the age of 18
* Patient must be able to give informed consent
* Women with child bearing potential must have a negative pregnancy test within seven days prior to the procedure

Exclusion Criteria:

* PaO2 less than 80 on FiO2 greater 70%
* Systolic blood pressure less than 90
* Active bronchospasm
* INR greater than 2.0 (INR: International Normalized Ratio)
* Recent myocardial infarction within last two weeks
* Active cardiac chest pain
* Significant untreated sleep apnea
* FEV1 less than 30% of predicted (FEV1: forced expiratory volume in 1 second)
* Worsening hypercarbia with PaCO2 greater than 55
* In active respiratory failure (unless endotracheal intubation is performed first to stabilize the airway)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-03 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Obtain biopsy correlated OFDI images with the purpose of establishing OFDI image criteria for discrimination of tissue types. | One time Bronchoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Carla R Lamb, M.D., Principal Investigator — Lahey Clinic, Inc.
Locations (1):
- Lahey Clinic, Inc., Burlington, Massachusetts, United States

REFERENCES:
- [Background] Jemal A, Siegel R, Ward E, Murray T, Xu J, Thun MJ. Cancer statistics, 2007. CA Cancer J Clin. 2007 Jan-Feb;57(1):43-66. doi: 10.3322/canjclin.57.1.43. PMID 17237035
- [Background] Society AC. Cancer Facts & Figures 2007. American Cancer Society. Atlanta, 2007
- [Background] Travis WD, Travis LB, Devesa SS. Lung cancer. Cancer. 1995 Jan 1;75(1 Suppl):191-202. doi: 10.1002/1097-0142(19950101)75:1+3.0.co;2-y. PMID 8000996
- [Background] Kerr KM. Pulmonary preinvasive neoplasia. J Clin Pathol. 2001 Apr;54(4):257-71. doi: 10.1136/jcp.54.4.257. PMID 11304841
- [Background] Hirsch FR, Franklin WA, Gazdar AF, Bunn PA Jr. Early detection of lung cancer: clinical perspectives of recent advances in biology and radiology. Clin Cancer Res. 2001 Jan;7(1):5-22. PMID 11205917
- [Background] Feller-Kopman D, Lunn W, Ernst A. Autofluorescence bronchoscopy and endobronchial ultrasound: a practical review. Ann Thorac Surg. 2005 Dec;80(6):2395-401. doi: 10.1016/j.athoracsur.2005.04.084. PMID 16305928
- [Background] Mountain CF. Revisions in the International System for Staging Lung Cancer. Chest. 1997 Jun;111(6):1710-7. doi: 10.1378/chest.111.6.1710. PMID 9187198
- [Background] Thiberville L. Nonsurgical therapeutic approach of early lung cancers of the proximal bronchus. European Respiratory Review 2002;12:182-186
- [Background] Sutedja TG, Schreurs AJ, Vanderschueren RG, Kwa B, vd Werf TS, Postmus PE. Bronchoscopic therapy in patients with intraluminal typical bronchial carcinoid. Chest. 1995 Feb;107(2):556-8. doi: 10.1378/chest.107.2.556. PMID 7842794
- [Background] Sato M, Saito Y, Endo C, Sakurada A, Feller-Kopman D, Ernst A, Kondo T. The natural history of radiographically occult bronchogenic squamous cell carcinoma: a retrospective study of overdiagnosis bias. Chest. 2004 Jul;126(1):108-13. doi: 10.1378/chest.126.1.108. PMID 15249450